CLINICAL TRIAL: NCT04592185
Title: Post-registration Observational Study on the Custom-made Abdominal Aortic Endograft Fenestrated Anaconda™
Brief Title: The Study of the Fenestrated Anaconda Device in the Treatment of Abdominal Aortic Aneurysms
Acronym: EPI-EFA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Vascutek Ltd. (Industry)
Collaborators: Federation of Medical Specialties (Other)
Responsible Party: Sponsor
Other Study IDs: EPI-EFA
Record Dates: First submitted 2020-10-15; First posted 2020-10-19 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Vascular Diseases; Aneurysm
Keywords: FEVAR; Fenestrated; Endovascular; AAA; Custom device
MeSH Terms: conditions — Vascular Diseases; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Fenestrated Anaconda™ Device — Treatment of complex abdominal aortic aneurysms

SUMMARY:
The French Ministry registered the Fenestrated Anaconda ™ on the List of Reimbursable Products and Services (LPPR) by the French Health Insurance on February 2018 for a duration of 5 years, while taking up the conditions for carrying out the act recommended by the CNEDiMTS (Committee in charge of medical device review), namely the carrying out of a post-registration study for the renewal of the authorization. This renewal of registration is conditioned by the set-up of a long-term follow-up study of all patients treated with the Fenestrated Anaconda ™ in France.

To do this, this study will be carried out in partnership with the Federation of Medical Specialties (FSM) and the National Professional Council (CNP) of Vascular Surgery in order to have the data necessary for the renewal of the registration of the Fenestrated Anaconda ™ from the registry called Datavasc developed by the CNP and available online on the FSM's electronic platform.

DETAILED DESCRIPTION:
EPI-EFA study: Post-registration study of the Fenestrated Anaconda™ in the management of a complex abdominal, juxtarenal, pararenal, suprarenal aortic aneurysm, whether or not associated with a distal common iliac artery or thoracoabdominal aneurysm type IV, in high-risk patients requiring treatment, for whom a surgical contraindication has been asked.

* Study type : observational, national, multi-centre, prospective, non-comparative study, as open registry
* Primary objective : To evaluate the long-term interest of Fenestrated Anaconda™ on all patients treated with in France. The data collected should be:
* 1-year mortality rate related to device, procedure, any cause = primary endpoint
* Stent-related adverse events (endoleak, migration, integrity of the device), renal events, ischemia (medullary (paraplegia / paraparesis), intestinal) = secondary endpoints
* Study timelines :
* Duration / follow-up :
* 1-year recruitment period from October 2019, with a minimum of 91 patients
* Mid-term follow-up : at 1 year
* Routine practice : until 5 years
* Reports to be submitted to French Health Authority :
* Interim report with mid-term follow-up data for renewal dossier
* Final report with long-term follow-up data

ELIGIBILITY:
At the request of the French Health Authority (HAS), no inclusion or exclusion criteria can be set as the study should be carried out on all patients treated with the device in France.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In order to meet the French Health Authority (HAS) requirements, this study aims to include all patients treated with the Fenestrated Anaconda™ under real conditions of use in France.
  These patients must have a preoperative morphological assessment favourable to the placement of a fenestrated endoprosthesis. The affected patients are considered at high risk.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Long-term outcome of use of Fenestrated Anaconda | 1 year
  Device-related mortality, procedure-related mortality, all-cause mortality

SECONDARY OUTCOMES:
Stent-related adverse events | 5 years
  Endoleak, migration, integrity of device
Renal adverse events | 5 years
  Renal adverse events
Ischemia | 5 years
  Medullary (paraplegia/paraparesis), intestinal

CONTACTS AND LOCATIONS:
Overall Officials: Pr. Jean-Noël Albertini, Principal Investigator — CHU de ST-ETIENNE- Hôpital Nord, SAINT-PRIEST-EN-JAREZ
Locations (33):
- France (33):
  - CHR de METZ-THIONVILLE - Hôpital de Mercy, Ars-Laquenexy
  - Clinique Belharra - BAYONNE, Bayonne
  - Clinique Saint-Vincent, Besançon
  - CHU de BESANCON, Besançon
  - Hôpital Privé de BOIS-BERNARD, Bois-Bernard
  - Clinique Saint-Augustin, Bordeaux
  - CHU de BORDEAUX - GH Pellegrin, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Clinique Convert de BOURG-EN-BRESSE, Bourg-en-Bresse
  - CHU de BREST - CH La Cavale Blanche, Brest
  - HCL - Hôpital L. Pradel - BRON, Bron
  - CHU de CLERMONT-FERRAND - site Gabriel-Montpied, Clermont-Ferrand
  - CHU de de DIJON BOURGOGNE - Hôpital François Mitterrand, Dijon
  - Clinique La Ligne Bleue, Épinal
  - Groupe Hospitalier Mutualiste de GRENOBLE, Grenoble
  - Centre Hospitalier d'ARCACHON, La Teste-de-Buch
  - APHM - Hôpital de La Timone, Marseille
  - APHM - Hôpital Nord, Marseille
  - Polyclinique Inkermann, Niort
  - Clinique Geoffroy St-Hilaire, Paris
  - Groupe Hospitalier Pitié-Salpêtrière, Paris
  - CH de PAU, Pau
  - CHU de BORDEAUX - Hôpital Haut-Lévêque, Pessac
  - CHU de REIMS - Hôpital Robert Debré, Reims
  - Clinique Mutualiste, Saint-Etienne
  - Clinique Belledonne, Saint-Martin-d'Hères
  - CHU de ST-ETIENNE- Hôpital Nord, Saint-Priest-en-Jarez
  - HU de STRASBOURG - Nouvel Hôpital Civil, Strasbourg
  - Polyclinique de l'Ormeau, Tarbes
  - CHU de NANCY - Hôpitaux de Brabois, Vandœuvre-lès-Nancy
  - Hôpital Robert Schuman, Vantoux
  - Hôpital Privé de VILLENEUVE D'ASCQ, Villeneuve-d'Ascq
  - Médipôle LYON-VILLEURBANNE, Villeurbanne

IPD SHARING:
Plan to Share IPD: No